CLINICAL TRIAL: NCT03415451
Title: Explore the Efficiency of Fiberscope-guided Nasogastric Tube Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201705078RIND
Record Dates: First submitted 2017-10-01; First posted 2018-01-30 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2018-12

CONDITIONS: Nasogastric Tube Esophagitis
Keywords: cancer patients, Nutritional status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fiberscope-Guided Nasogastric tube (Experimental): Fiberscope-Guided Nasogastric tube insertion
  Interventions: Device: Fiberscope-Guided Nasogastric tube insertion

INTERVENTIONS:
Device: Fiberscope-Guided Nasogastric tube insertion — Fiberscope-Guided Nasogastric tube insertion

SUMMARY:
For Head and neck cancer and uncooperative patients, blind nasogastric tube (NGT) insertion may sometimes be very difficult because of the anatomical obstructions in the pharynx and uncoordinated swallowing motion. To solve the problem, flexible endoscope has been used widely to assist the NGT insertion via direct visual assistance, working channels/guide wires, or suture fixation. Unfortunately, these tools are not easily assessed in the outpatient department. Here, we try to use a simpler method for the flexible endoscope to guide the NGT insertion.

DETAILED DESCRIPTION:
NGT and fiberscope was combined to facilitate NG tube insertion

ELIGIBILITY:
Inclusion criteria: dysphagia patients who need nasogastric tube feeding Exclusion criteria: Patients who ever had human immunodeficiency virus infection and were not suitable for fiberscope exam without protection sheath

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
The success rates of fiberscope-guided NG tube insertion | 1 year
  fiberscope-guided NG tube insertion

CONTACTS AND LOCATIONS:
Overall Officials: CHI-MAW LIN, MD, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan